CLINICAL TRIAL: NCT01175590
Title: A Study to Evaluate the Safety of Besivance™ (Besifloxacin Ophthalmic Suspension) 0.6% Compared to Vehicle Following Three Times Daily(TID) Dosing for 7 Days
Brief Title: Safety of Besivance™ (Besifloxacin Ophthalmic Suspension) 0.6% Compared to Vehicle
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 631
Record Dates: First submitted 2010-08-03; First posted 2010-08-05 (Estimated); Results first posted 2013-05-01 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-03

CONDITIONS: Bacterial Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Bacterial | interventions — besifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Besivance (Experimental): besifloxacin ophthalmic suspension 0.6%
  Interventions: Drug: Besivance
- Vehicle (Placebo Comparator): Vehicle of Besivance
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Besivance — Ocular administration to affected eye for 7 days
  Arms: Besivance
Drug: Vehicle — Vehicle of Besivance administered to affected eye for 7 days
  Arms: Vehicle

SUMMARY:
The objective of this study is to evaluate the safety of Besivance (besifloxacin ophthalmic suspension, 0.6%) compared to vehicle.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a clinical diagnosis of acute bacterial conjunctivitis and exhibit purulent conjunctival discharge (crusty or sticky eyelids) and redness in at least one eye.
* Subjects who are willing to discontinue contact lens wear for the duration of the study.
* Subjects who are able and willing to comply with all treatment and follow- up/study procedures.

Exclusion Criteria:

* Subjects who have any uncontrolled systemic disease or debilitating disease.
* Subjects with a known hypersensitivity or contraindications to Besivance, fluoroquinolones, or any of the ingredients in the study drugs.
* Subjects who are expected to require disallowed concurrent systemic or ocular therapy(either eye)during or prior to study start. (ie, NSAIDs, corticosteroids, mast cell stabilizers, antihistamines, decongestants or antimicrobial therapy)
* Subjects having ocular surgery (including laser surgery) in either eye within six weeks prior to entry into this study.
* Subjects with suspected viral or allergic conjunctivitis or any other disease conditions that could interfere with the efficacy and safety evaluations of the study medication.
* Subjects with suspected iritis.
* Subjects with a history of recurrent corneal erosion syndrome, either idiopathic or secondary to previous corneal trauma or dry eye syndrome.
* Subjects with any active ulcerative keratitis, specifically any epithelial loss greater than punctate keratitis.
* Subjects who are immune compromised.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Allaire, MD, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb, Inc., Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant entered the study 6/22/2010 and the last participant visit was 12/12/2011. Twenty four sites in the United States participated in the study.
Pre-assignment Details: 518 participants with a clinical diagnosis of bacterial conjunctivitis were enrolled in the study, 496 completed the study; 518 participants were in Intent-to-Treat (ITT) population, 514 participants were in Safety population, and 299 participants were in modified Intent-to-Treat (mITT) population (Participants with positive culture at baseline).
Groups:
- Besivance: besifloxacin ophthalmic suspension 0.6%
  Besivance : Ocular administration to affected eye for 7 days
- Vehicle: Vehicle of Besivance
  Vehicle : Vehicle of Besivance administered to affected eye for 7 days
Period: Overall Study
Arm/Group | Besivance | Vehicle
Started | 347 | 171
Modified Intent to Treat Population | 212 | 87
Safety Population | 344 | 170
Completed | 335 | 161
Not Completed | 12 | 10
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Adverse Event | 4 | 0
Not completed — Physician Decision | 1 | 4
Not completed — Lack of Efficacy | 1 | 1
Not completed — Residual Bacterial Conjunctivitis | 1 | 0
Not completed — Treated not as randomized | 3 | 2
Not completed — Herpes Simplex Dermatitis | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat population (ITT)
Groups:
- Total: Total of all reporting groups
Arm/Group | Besivance | Vehicle | Total
Number analyzed (Participants) | 347 | 171 | 518
Age, Customized [Number; unit: participants]
  0-17 years | 149 | 62 | 211
  18 - 49 years | 106 | 71 | 177
  >=50 years | 92 | 38 | 130
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 205 | 95 | 300
  Male | 142 | 76 | 218
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 3 | 10
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 83 | 40 | 123
  White | 213 | 103 | 316
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 39 | 19 | 58

OUTCOME MEASURES:

1. Primary Outcome: Ocular Treatment Emergent Adverse Events
Description: Ocular Treatment-Emergent Adverse Events on the Study Eye
Time Frame: At each visit - 7 days
Population: Safety Population
Measure: Number; unit: Events
Units Other Than Participants: eyes
Arm/Group | Besivance | Vehicle
Number analyzed (Participants) | 344 | 170
Number analyzed (eyes) | 344 | 170
Events
  Conjunctivitis | 3 [0.2 to 3] | 3 [0.4 to 5.1]
  Blepharitis | 1 [0.0 to 1.6] | 1 [0.0 to 3.2]
  Conjunctival Oedema | 1 [0.0 to 1.6] | 1 [0.0 to 3.2]
  Erythema of Eyelid | 2 [0.1 to 2.1] | 0 [0.0 to 0.0]
  Punctate Keratitis | 1 [0.0 to 1.6] | 1 [0.0 to 3.2]
  Conjunctival Haemorrhage | 1 [0.0 to 1.6] | 0 [0.0 to 0.0]
  Conjunctivitis Allergic | 0 [0.0 to 0.0] | 1 [0.0 to 3.2]
  Corneal Infiltrates | 1 [0.0 to 1.6] | 0 [0.0 to 0.0]
  Dacryocystitis | 1 [0.0 to 1.6] | 0 [0.0 to 0.0]
  Eye Pain | 1 [0.0 to 1.6] | 0 [0.0 to 0.0]
  Lacrimation Increased | 1 [0.0 to 1.6] | 0 [0.0 to 0.0]
  Scleritis | 0 [0.0 to 0.0] | 1 [0.0 to 3.2]
  Instillation Site Reaction | 2 [0.1 to 2.1] | 1 [0.0 to 3.2]
  Instillation Site Erythema | 1 [0.0 to 1.6] | 0 [0.0 to 0.0]
  Instillation Site Irritation | 0 [0.0 to 0.0] | 1 [0.0 to 3.2]
  Instillation Site Pain | 1 [0.0 to 1.6] | 0 [0.0 to 0.0]
  Pain | 0 [0.0 to 0.0] | 1 [0.0 to 3.2]
  Herpes Dermatitis | 1 [0.0 to 1.6] | 0 [0.0 to 0.0]
  Post-Traumatic Pain | 0 [0.0 to 0.0] | 1 [0.0 to 3.2]
  Corneal Staining | 1 [0.0 to 1.6] | 0 [0.0 to 0.0]

2. Secondary Outcome: Clinical Resolution
Description: The absence of both conjunctival discharge and bulbar conjunctival injection, after seven days of treatment. Participants with non-missing data
Time Frame: Day 8 (Visit 2)
Population: Study eye for the mITT population
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Besivance | Vehicle
Number analyzed (Participants) | 206 | 83
Number analyzed (eyes) | 206 | 83
eyes | 112 | 46

3. Secondary Outcome: Clinical Resolution
Description: The absence of both conjunctival discharge and bulbar conjunctival injection, after seven days of treatment.
Time Frame: Day 11 (Visit 3)
Population: Study eye for the mITT population
Measure: Number; unit: eyes
Arm/Group | Besivance | Vehicle
Number analyzed (Participants) | 204 | 84
eyes | 169 | 68

4. Secondary Outcome: Microbial Eradication
Description: The absence of all accepted ocular bacterial species that were present at or above threshold at baseline, after seven days of treatment.
Time Frame: Days 8 (Visit 2)
Population: Study Eye, Modified Intent-to-Treat Population
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Besivance | Vehicle
Number analyzed (Participants) | 206 | 80
Number analyzed (eyes) | 206 | 80
eyes | 172 | 36

5. Secondary Outcome: Microbial Eradication
Description: as for outcome 4
Time Frame: Days 11 (Visit 3)
Population: Study Eye, Modified Intent-to-Treat Population
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Besivance | Vehicle
Number analyzed (Participants) | 200 | 83
Number analyzed (eyes) | 200 | 83
eyes | 169 | 48

6. Primary Outcome: Non-Ocular Treatment-Emergent Adverse Events
Description: Non-Ocular Treatment-Emergent Adverse Events on the Study Eye
Time Frame: 7 days
Population: Safety Population
Measure: Number; unit: Events
Arm/Group | Besivance | Vehicle
Number analyzed (Participants) | 344 | 170
Events
  Ear Pain | 1 [0.0 to 1.6] | 0 [0.0 to 0.0]
  Dysgeusia | 1 [0.0 to 1.6] | 0 [0.0 to 0.0]
  Pyrexia | 1 [0.0 to 1.6] | 0 [0.0 to 0.0]
  Nasopharyngitis | 2 [0.1 to 2.1] | 1 [0.0 to 3.2]
  Bronchitis | 0 [0.0 to 0.0] | 1 [0.0 to 3.2]
  Gastroenteritis, Viral | 0 [0.0 to 0.0] | 1 [0.0 to 3.2]
  Otitis Media | 1 [0.0 to 1.6] | 0 [0.0 to 0.0]
  Upper Respiratory Tract Infection | 1 [0.0 to 1.6] | 0 [0.0 to 0.0]

7. Secondary Outcome: Microbial Outcome With Clinical Resolution
Description: At each follow-up visit for the accepted ocular bacterial species that were present at or above threshold at baseline
Time Frame: Day 8 (Visit 2)
Population: Modified Intent-to-Treat Population
Measure: Number; unit: eyes
Arm/Group | Besivance | Vehicle
Number analyzed (Participants) | 206 | 80
eyes
  Clinical Resolution with Microbial Eradication | 96 | 22
  Clinical Resolution with no Microbial Eradication | 16 | 24
  No Clinical Resolution with Microbial Eradication | 76 | 14
  No Clinical Resolution no Microbial Eradication | 18 | 20

8. Secondary Outcome: Microbial Outcome With Clinical Resolution
Description: At each follow-up visit for the accepted ocular bacterial species that were present at or above threshold at baseline
Time Frame: Day 11 (Visit 3)
Population: Modified Intent-to-Treat Population
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Besivance | Vehicle
Number analyzed (Participants) | 200 | 83
Number analyzed (eyes) | 200 | 83
eyes
  Clinical Resolution with Microbial Eradication | 143 | 42
  Clinical Resolution with no Microbial Eradication | 23 | 25
  No Clinical Resolution with Microbial Eradication | 26 | 6
  No Clinical Resolution no Microbial Eradication | 8 | 10

9. Secondary Outcome: Individual Clinical Outcomes - Ocular Discharge
Description: ocular conjunctival discharge measured as absent, mild, moderate or severe
Time Frame: At day 1 (Vist 1)
Population: Baseline-Designated Study Eye (Modified Intent-to- Treat Population)
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Besivance | Vehicle
Number analyzed (Participants) | 212 | 87
Number analyzed (eyes) | 212 | 87
eyes
  Absent | 0 | 0
  Mild | 94 | 38
  Moderate | 106 | 44
  Severe | 12 | 5

10. Secondary Outcome: Individual Clinical Outcomes - Ocular Discharge
Description: ocular conjunctival discharge measured as absent, mild, moderate or severe
Time Frame: At day 8 (Vist 2)
Population: Baseline-Designated Study Eye (Modified Intent-to- Treat Population)
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Besivance | Vehicle
Number analyzed (Participants) | 206 | 83
Number analyzed (eyes) | 206 | 83
eyes
  Absent | 155 | 61
  Mild | 42 | 18
  Moderate | 8 | 4
  Severe | 1 | 0

11. Secondary Outcome: Individual Clinical Outcomes - Ocular Discharge
Description: ocular conjunctival discharge measured as absent, mild, moderate or severe
Time Frame: At day 11 (Vist 3)
Population: Baseline-Designated Study Eye (Modified Intent-to- Treat Population)
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Besivance | Vehicle
Number analyzed (Participants) | 204 | 84
Number analyzed (eyes) | 204 | 84
eyes
  Absent | 187 | 77
  Mild | 12 | 6
  Moderate | 4 | 1
  Severe | 1 | 0

12. Secondary Outcome: Individual Clinical Outcomes - Bulbar Injection
Description: Bulbar conjunctival injection measured as normal, mild, moderate or severe
Time Frame: At day 1 (Vist 1)
Population: Baseline-Designated Study Eye (Modified Intent-to- Treat Population)
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Besivance | Vehicle
Number analyzed (Participants) | 212 | 87
Number analyzed (eyes) | 212 | 87
eyes
  Normal | 0 | 0
  Mild | 110 | 44
  Moderate | 83 | 37
  Severe | 19 | 6

13. Secondary Outcome: Individual Clinical Outcomes - Bulbar Injection
Description: Bulbar conjunctival injection measured as normal, mild, moderate or severe
Time Frame: At day 8 (Vist 2)
Population: Baseline-Designated Study Eye (Modified Intent-to- Treat Population)
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Besivance | Vehicle
Number analyzed (Participants) | 206 | 83
Number analyzed (eyes) | 206 | 83
eyes
  Normal | 142 | 57
  Mild | 56 | 23
  Moderate | 7 | 3
  Severe | 1 | 0

14. Secondary Outcome: Individual Clinical Outcomes - Bulbar Injection
Description: Bulbar conjunctival injection measured as normal, mild, moderate or severe
Time Frame: At day 11 (Vist 3)
Population: Baseline-Designated Study Eye (Modified Intent-to- Treat Population)
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Besivance | Vehicle
Number analyzed (Participants) | 204 | 84
Number analyzed (eyes) | 204 | 84
eyes
  Normal | 182 | 72
  Mild | 18 | 11
  Moderate | 4 | 1
  Severe | 0 | 0

ADVERSE EVENTS:
Time Frame: 11 days
Arm/Group | Besivance | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/347 | 0/171
Other Adverse Events (participants affected / at risk) | 0/347 | 0/171

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed. Prior to publication or presentation, a copy of the final text should be forwarded by the Investigator(s) to the Sponsor or its designee, for comment.